CLINICAL TRIAL: NCT05969873
Title: Effect Of Pilates On Postural Control And Balance In Children With Down's Syndrome
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Riphah International University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: REC/RCR & AHS/23/0727
Record Dates: First submitted 2023-07-23; First posted 2023-08-01 (Actual); Last update posted 2023-12-27 (Actual); Status verified 2023-12

CONDITIONS: Down Syndrome
Keywords: Balance; Contrology; Down syndrome; Pilates; Pediatric Balance Scale
MeSH Terms: conditions — Down Syndrome | interventions — Exercise Movement Techniques; Control Groups

STUDY DESIGN:
Intervention Model Description: The study will be randomized controlled trial used to evaluate the effectiveness of pilates on posture and balance in children with down's syndrome. Subjects with down's syndrome meeting the pre-detremined inclusion and exclusion criteria will be divided into two groups using non-probability sampling technique.
Who Masked: Participant
Masking Description: Participants will get separate treatment protocols and possible efforts will be put to mask the both groups about their treatment.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Pilates Group (Experimental): In this group patients will be treated with physical therapy treatment pilates exercise. Group A underwent 45 minutes of Pilates exercises in addition to the identical exercise programme as group A to improve the strength, coordination and flexibility of the lower limbs. Pilates movements were carried out ten times, with a two-minute break in between each repetition. For six weeks, both groups participated in the intervention programme three times per week. Starting the programme off with supine exercises of segmental motions that include using the trunk muscles to maintain a neutral posture is normal. To enhance shoulder girdle control, supine arm workouts were gradually added. The spine's ability to flex and extend was steadily increased.
  Interventions: Other: Pilates exercise
- Balance training group (Active Comparator): In this group patients will be treated with PT treatment with balance training. Exercises for stability of posture on numerous surfaces and positions were performed by Group B, including exercises for the flexors and adductors of hip, flexors and extensors of knee, and calf muscle (15-second hold and five repetitions) for improving their flexibility. The lower extremity and trunk muscles were the focus of Group B. The postural control exercise included walking in every direction, moving past the point of stability in various postures like half-kneeling, standing on hard and soft surfaces, stepping down and up, walking and standing at the same time, and one leg standing with eyes open and closed. Each session started with a 5-minute warm-up and ended with a 5-minute cool-down in between each phase.
  Interventions: Other: Balance training

INTERVENTIONS:
Other: Pilates exercise — Patients in this group will be treated with pilates exercise and conventional physical therapy as baseline treatment.
  Other Names: Experimental group
  Arms: Pilates Group
Other: Balance training — Patients in this group will be treated with balance training and conventional physical therapy as baseline treatment.
  Other Names: Control group
  Arms: Balance training group

SUMMARY:
Down's syndrome (DS) is a genetic condition characterized by the presence of an extra chromosome 21, leading to various clinical symptoms. Individuals with DS often experience challenges in balance, posture, and motor skills, which can impact their daily activities. Pilates activities focus on the concept of control of muscles. Pilates increases trunk flexibility, abdominal and core strength and endurance, and deep core muscle activation hence improving balance and posture.

DETAILED DESCRIPTION:
The study will be randomized controlled trial used to evaluate the effectiveness of pilates on posture and balance in children with down's syndrome. Subjects with down's syndrome meeting the pre-detremined inclusion and exclusion criteria will be divided into two groups using non-probability sampling technique. Assessment will be done using Pediatric balance scale(PBS) and Timed up and go test (TUG).). Control group will receive regular physical therapy with balance training and experimental group will receive regular physical therapy+ Pilates.

ELIGIBILITY:
Inclusion Criteria:

* Down's syndrome children with age between 6 and 12 years.
* The ability to execute required motor skill proficiency and executive function tests.
* The capacity to walk and stand by oneself

Exclusion Criteria:

* • Children who are not able to comprehend commands.

  * Associated cardiovascular and orthopedic condition.
  * Loss of functional hearing and vision or a related respiratory disease.
  * History of traumatic injury
  * History of previous surgery
  * Inability of parents to understand the procedure and their unwillingness to participate

Ages: 6 Years to 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 22 (Actual)
Dates: Start 2023-07-16 (Actual); Primary Completion 2023-11-01 (Actual); Study Completion 2023-11-15 (Actual)

PRIMARY OUTCOMES:
Pediatric Balance Scale | 12 weeks
  This tool is used for assessing change from baseline. The PBBS is easy to administer, does not require specialized equipment, and can be completed in <20 minutes. A 0 to 4 grading scale provides a quantitative and qualitative measure of performance. It involves 14 mobility tasks, with the tasks varying in degrees of difficulty. The tasks are divided into 3 domains: sitting balance, standing balance, and dynamic balance. PBS has high validity and reliability of 0.98. 41-56= low fall risk, 21-40= medium fall risk, 0-20=high risk

SECONDARY OUTCOMES:
Timed up and go test | 12 weeks
  TUG is a simple test used to assess a person's mobility and evaluate both static and dynamic balance. It uses the time that a person takes to rise from a chair, walk three meters, turns around 180 degrees, walk back to the chair and sit down while turning 180 degrees.
  Interpretation: ≤ 10 seconds= normal. A score of ≥ 14 seconds has been shown to indicate high risk of fall.
  ICC value for interrater reliability between 2 authors' TUG times for 20 randomly selected patients was .96.

CONTACTS AND LOCATIONS:
Overall Officials: Rida Khawar Dar, MS*, Principal Investigator — Riphah International University
Locations (1):
- Riphah International University, Lahore, Punjab Province, Pakistan

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Abd-Elfattah HM, Galal DOSM, Aly MIE, Aly SM, Elnegamy TE. Effect of Pilates Exercises on Standing, Walking, and Balance in Children With Diplegic Cerebral Palsy. Ann Rehabil Med. 2022 Feb;46(1):45-52. doi: 10.5535/arm.21148. Epub 2022 Feb 28. PMID 35272439